CLINICAL TRIAL: NCT05939635
Title: Bilateral Ultrasound-guided M-Tapa Block vs External Oblique Intercostal Block for Postoperative Analgesia in Patients Undergoing Laparoscopic Sleeve Gastrectomy Surgery: A Prospective Randomized Controlled Study
Brief Title: M-Tapa Block vs External Oblique Intercostal Block for Laparoscopic Sleeve Gastrectomy Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, BURHAN DOST, Associate Professor, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MTAPAEOIBLSG2023
Record Dates: First submitted 2023-06-23; First posted 2023-07-11 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Anesthesia; Regional Anesthesia; Postoperative Pain
Keywords: Anesthesia; Nerve block; Sleeve gastrectomy; External oblique intercostal block
MeSH Terms: conditions — Pain, Postoperative | interventions — Dental Occlusion

STUDY DESIGN:
Intervention Model Description: A block randomization list will be created by a doctor who does not participate in patient follow-up using a web-based program.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Researchers, surgeons and nurses, and those involved in study outcome analysis will not be aware of the randomization of the group. Block quality and standardization will be performed by an anesthetist experienced in regional anesthesia for EOIB and M-TAPA block.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group M-TAPA (Active Comparator): A bilateral M-TAPA (60 ml, %0.25 bupivacaine, totally) + IV morphine patient-controlled analgesia (PCA)
  Interventions: Procedure: Bilateral ultrasound guided Modified thoracoabdominal nerves block through perichondrial approach(M-TAPA) block; Drug: IV morphine patient-controlled analgesia (PCA)
- Group EOIB (Active Comparator): A bilateral EOIB (60 ml, %0.25 bupivacaine, totally) + IV morphine patient-controlled analgesia (PCA)
  Interventions: Procedure: Bilateral ultrasound guided external oblique intercostal block (EOIB); Drug: IV morphine patient-controlled analgesia (PCA)

INTERVENTIONS:
Procedure: Bilateral ultrasound guided external oblique intercostal block (EOIB) — Bilateral ultrasound-guided EOIB (total of 60 ml, %0.25 bupivacaine) will be performed + IV morphine PCA Multimodal analgesia : Patients are administered iv tenoxicam 20mg and tramadol 100 mg after induction of general anesthesia, and iv paracetamol 1 gr and 0.05 mg/kg, ideal body weight (IBW), iv morphine will be administered. End of the surgery, hyoscine-N-butyl bromide will be administered. Postoperative analgesia: iv paracetamol 1gr every 8 hours and IV PCA of 0,5 mg/ml morphine (the bolus dose is 20 μg/kg, the lock-in time of 6-10 minutes, the 4-hour limit is adjusted to be 80% of the calculated total amount). In cases where rescue analgesia is required (NRS score ≥4), 50 mg of meperidine is administered to patients.
  Patients are routinely administered ondansetron 8 mg IV 20 minutes before extubation for postoperative nausea and vomiting prophylaxis.
  Other Names: External oblique intercostal block (EOIB)
  Arms: Group EOIB
Procedure: Bilateral ultrasound guided Modified thoracoabdominal nerves block through perichondrial approach(M-TAPA) block — Bilateral ultrasound guided Modified thoracoabdominal nerves block through perichondrial approach(M-TAPA) block (total of 60 ml, %0.25 bupivacaine) will be performed + IV morphine PCA Multimodal analgesia : Patients are administered iv tenoxicam 20mg and tramadol 100 mg after induction of general anesthesia, and iv paracetamol 1 gr and 0.05 mg/kg, ideal body weight (IBW), iv morphine will be administered. End of the surgery, hyoscine-N-butyl bromide will be administered. Postoperative analgesia: iv paracetamol 1gr every 8 hours and IV PCA of 0,5 mg/ml morphine (the bolus dose is 20 μg/kg, the lock-in time of 6-10 minutes, the 4-hour limit is adjusted to be 80% of the calculated total amount). In cases where rescue analgesia is required (NRS score ≥4), 50 mg of meperidine is administered to patients.
  Patients are routinely administered ondansetron 8 mg IV 20 minutes before extubation for postoperative nausea and vomiting prophylaxis.
  Other Names: M-TAPA block
  Arms: Group M-TAPA
Drug: IV morphine patient-controlled analgesia (PCA) — Morphine will be administered via PCA device for the first 24 hours after surgery
  Other Names: morphine PCA

SUMMARY:
In obese patients, adequate pain relief in the postoperative period is an important parameter that affects patient comfort and hospital stay. Increasing patient comfort and recovery quality can be achieved by avoiding undesirable effects such as nausea, vomiting, and analgesia. This study aimed to investigate the effects of Bilateral External Oblique Intercostal Block (EOIB) and Perichondrial Modified Thoracoabdominal Nerve Block (M-TAPA) on postoperative acute pain scores (0-24 hours) and 24-hour opioid consumption in patients who underwent laparoscopic sleeve gastrectomy.

DETAILED DESCRIPTION:
Morbid obesity patients often have multisystem physiological changes and multiple comorbidities that can significantly affect perioperative pain control. These patients may have increased side effects from inadequate acute pain management and opioids should be used with caution.

Regional techniques can be applied in obese patients because they provide non-opioid analgesia and have fewer perioperative respiratory side effects. Effective pain control is associated with reduced post-operative opioid administration, faster mobilization, faster recovery, and shorter hospital stay.

Intraoperative nerve blocks using local anesthetics have been shown to improve postoperative pain in various abdominal surgeries, both open and laparoscopic. Recently, it has been reported that the M-TAPA block is a promising new technique that provides effective analgesia of the anterior and lateral thoracoabdominal walls during laparoscopic surgery, in which local anesthetic is delivered only to the underside of the perichondral surface.

TAPA/M-TAPA block has been shown to provide a potent analgesic effect in a large abdomen by numbing both the anterior and lateral cutaneous branches of the thoracoabdominal nerves. Therefore, the TAPA/M-TAPA block has been used in various abdominal surgeries. The EOI block represents an important modification of the fascial plane block techniques that can consistently cover the upper lateral abdominal wall.

When we look at the literature, it is seen that there are not enough studies on M-TAPA block and EOIB.

The aim of this study is to investigate the effects of Bilateral External Oblique Intercostal Block (EOIB) and Perichondrial Modified Thoracoabdominal Nerve Block (M-TAPA) on postoperative acute pain scores (0-24 hours) and 24-hour opioid consumption in patients who underwent laparoscopic sleeve gastrectomy. Our study, which the investigators think will contribute to the literature, was planned as a prospective, randomized, controlled, parallel-group study.

Patients will be divided into two groups:

Group M-TAPA :

A bilateral M-TAPA (60 ml 0.25% bupivacaine + 1:400.000 adrenaline) will be performed. In addition, IV morphine-PCA will be applied postoperatively for 24 hours.

Group EOIB :

A bilateral EOIB (60 ml 0.25% bupivacaine + 1:400.000 adrenaline) will be performed. In addition, IV morphine-PCA will be applied postoperatively for 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* Age between18-65 years
* American Society of Anesthesiology score II-III
* Body mass index (BMI) > 35 kg/m2
* Patients who will sign the informed consent form

Exclusion Criteria:

* History of opioid use for more than four weeks
* Chronic pain syndromes
* Patients with a history of local anesthetic or opioid allergy, hypersensitivity
* Severe cardiac, hepatic, and renal disease
* Alcohol and drug addiction
* Conditions where regional anesthesia is contraindicated
* Failure in the dermatomal examination performed after the block
* Patients with a STOP-BANG score ≥5

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2023-07-11 (Actual); Primary Completion 2023-10-26 (Actual); Study Completion 2024-01-29 (Actual)

PRIMARY OUTCOMES:
Morphine consumption in the first 24 hours after surgery | Postoperative day 1
  Morphine consumption in the first 24 hours after surgery will be measured. Patients can request opioids via a PCA device when their NRS score is≥ 4.

SECONDARY OUTCOMES:
Postoperative pain scores | Postoperative day 1
  Pain status at rest and while activity will be assessed by NRS score at 0, 3, 6, 12, 18, and 24 hours after surgery. The NRS is an 11-point numeric scale that ranges from 0 to 10.
Patients' satisfaction and quality of pain management | Postoperative day 1
  Patients' pain management satisfaction and quality will be evaluated using the QoR-15 score. The QoR-15 consists of 5 test areas: pain (2 questions), physical comfort (5 questions), physical state (2 questions), psychological state (2 questions), and emotional state (4 questions). Each question is rated on a 10-point scale ranging from 0 = "never" to 10 = "always" (scoring is reversed for negative questions).
  QoR-15 Turkish Version will be used for assessment.
The incidences of postoperative nausea and vomiting (PONV) | Postoperative day 1
  The severity of postoperative nausea and vomiting (PONV) will be assessed using a descriptive verbal rating scale at 0, 3, 6, 12, 18, and 24 hours after extubation. If a score of 3 or more, ondansetron 4 mg IV will be administered and will repeat after 8 hours if required. The PONV scale is 0 = no nausea; 1 = slight nausea; 2 = moderate nausea; 3 = vomiting once; and 4 = vomiting more than once.
Time of first analgesic request | Postoperative day 1
  Time at which the first analgesic is requested
Intraoperative remifentanil consumption | The remifentanil consumption will be recorded from anesthesia induction until the patient is referred to the recovery unit, up to 150 minutes.
  The total amount of remifentanil consumed will be recorded.
The number of patients with complications | Postoperative 7 days on an average
  The number of patients has any complications -directly related to the block or the drug used in the block- will be recorded
The number of patients who required rescue analgesia. | Postoperative day 1
  he number of patients requiring rescue analgesics will be recorded over 24 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Burhan DOST, Md, Study Director — Ondokuz Mayıs University Faculty of Medicine
Locations (1):
- Ondokuz Mayis University, Samsun, Atakum, Turkey (Türkiye)

REFERENCES:
- [Background] Gungor H, Ciftci B, Alver S, Golboyu BE, Ozdenkaya Y, Tulgar S. Modified thoracoabdominal nerve block through perichondrial approach (M-TAPA) vs local infiltration for pain management after laparoscopic cholecystectomy surgery: a randomized study. J Anesth. 2023 Apr;37(2):254-260. doi: 10.1007/s00540-022-03158-0. Epub 2022 Dec 28. PMID 36575362
- [Background] White L, Ji A. External oblique intercostal plane block for upper abdominal surgery: use in obese patients. Br J Anaesth. 2022 May;128(5):e295-e297. doi: 10.1016/j.bja.2022.02.011. Epub 2022 Mar 3. No abstract available. PMID 35249704
- [Background] Erskine RN, White L. "A review of the external oblique intercostal plane block - a novel approach to analgesia for upper abdominal surgery". J Clin Anesth. 2022 Nov;82:110953. doi: 10.1016/j.jclinane.2022.110953. Epub 2022 Aug 19. No abstract available. PMID 35994942
- [Background] Ibrahim M, Elnabtity AM, Hegab A, Alnujaidi OA, El Sanea O. Combined opioid free and loco-regional anaesthesia enhances the quality of recovery in sleeve gastrectomy done under ERAS protocol: a randomized controlled trial. BMC Anesthesiol. 2022 Jan 21;22(1):29. doi: 10.1186/s12871-021-01561-w. PMID 35062872